CLINICAL TRIAL: NCT03618121
Title: Innovations in Biofeedback and Its Use in Mental Health
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Primary Investigator is leaving host university (ETSU)
Sponsor: East Tennessee State University (Other)
Responsible Party: Principal Investigator, Jason Steadman, Assistant Professor of Psychology, East Tennessee State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0516.15f
Record Dates: First submitted 2018-07-23; First posted 2018-08-07 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Anxiety; Biofeedback, Psychology
Keywords: Videogames; Commercial biofeedback device
MeSH Terms: conditions — Anxiety Disorders | interventions — Biofeedback, Psychology; Relaxation Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Biofeedback plus gaming (Nevermind) (Experimental): 1) Group A is a biofeedback plus gaming group. Participants in this group play a horror videogame called Nevermind, while also wearing a chest strap heart rate monitor. The object of the videogame is to assist a patient by entering his/her mind and helping him/her work through some trauma memories. The way the game works is that the more anxious players are, the faster their heart beats, and the faster the heart beats, the harder and scarier the game gets. Thus, in order for one to do well in the game, he or she has to learn how to control the heartbeat and stress through relaxation. A therapist will help people in this group to learn relaxation techniques to help calm their body and finish the game.
  Interventions: Device: Biofeedback plus gaming (Nevermind)
- Gaming only (Active Comparator): 2) Group B is a gaming only group. Like Group A, participants in this group play a Nevermind, but this time they do not wear a heart rate monitor. A therapist will still be present to help people in this group to learn relaxation techniques to help calm themselves during game play, but in this case the game does not change based on heart rate.
  Interventions: Behavioral: Gaming only
- Biofeedback only (The Pip) (Active Comparator): 3) Group C is a biofeedback only group. In Group C, participants use a device called The Pip that measures Galvanic Skin Response. The Pip interacts with a few basic apps used in this study to teach relaxation. In one app, players control flying dragons. The more relaxed players are (as measured by GSR), the higher and faster their dragon flies. In another app, players control the changing of seasons. The more relaxed players are, the faster they can make seasons change from winter to spring. In another app, players can watch a simple graph of their stress over a period of time. Participants can learn to decrease stress by learning to make the line on the graph go down. In Group C, a therapist will also be present with participants to help them learn techniques to reduce stress.
  Interventions: Device: Biofeedback only (The Pip)
- Relaxation training only (Active Comparator): 4) Group D is a relaxation training only group. In Group D, participants receive relaxation training from a trained therapist. Participants in this group learn and practice with their therapist different techniques to help them relax and reduce stress.
  Interventions: Behavioral: Relaxation training

INTERVENTIONS:
Device: Biofeedback plus gaming (Nevermind) — Participants will receive relaxation training from a trained therapist while receiving biofeedback through the game Nevermind. Participants receive two 30-minute sessions per week, for 4 weeks, for a total of 8 sessions.
  Arms: Biofeedback plus gaming (Nevermind)
Device: Biofeedback only (The Pip) — Participants receive relaxation training from a trained therapist with biofeedack through The Pip device. The Pip connects with 4 apps, The Loom, Relax & Race, PipStressTracker, and Clarity. All 4 will be used in this study. Participants receive 2 30-minute sessions per week, for 4 weeks, for a total of 8 sessions.
  Arms: Biofeedback only (The Pip)
Behavioral: Relaxation training — Standard relaxation training protocol often used in clinical care. Participants receive 2 30-minute sessions per week, for 4 weeks, for a total of 8 sessions.
  Arms: Relaxation training only
Behavioral: Gaming only — Intervention is identical to the "Biofeedback plus gaming (Nevermind)" intervention, but in this case participants play Nevermind without any biofeedback. Thus, they receive 2 30-minute sessions of relaxation training per week, for 4 weeks, totaling 8 sessions. During relaxation training, they will play the Nevermind game, but without attaching to any biofeedback devices.
  Arms: Gaming only

SUMMARY:
This study investigates the use of new technologies in "biofeedback gaming" and their potential for use as a treatment for stress and anxiety. Biofeedback training is typically accomplished through devices that measure heartrate variability (HRV), galvanic skin response (GSR), or electroencephalogram (EEG). Typically, the use of this equipment requires a practitioner with specialized training in reading and interpreting HRV, GSR, and/or EEG. However, recent advances in technology have made biofeedback devices more readily available to the general public, and some commercial devices are now being sold. This study investigates the utility of these commercial devices with a mild clinical population. In this study, participants use two tools for biofeedback training, one is called "The Pip," described in Group C, below, and another is a computer game called Nevermind, described in Groups A and B, below. These are compared against a control group (group D), which is standard relaxation training without biofeedback.

ELIGIBILITY:
Inclusion criteria:

1. Participant scores at least 1.5 standard deviations above the mean on any anxiety or stress-based scale (BAI or PSS), OR
2. Patient is assigned a CSR of 4 or higher on any anxiety disorder using the ADIS-5, OR
3. Patient exhibits maladaptive coping strategies, as demonstrated by COPE profile, AND
4. Patient shows some level of functional impairment as a result of stress, anxiety, and/or restlessness (i.e. the symptoms are judged by clinician to be clinically meaningful).

Exclusion criteria:

1. Participant is not English-speaking.
2. Participant appears to meet criteria for a comorbid psychiatric diagnosis that warrants alternative psychological treatment (e.g. PTSD, OCD, Major Mood Disorder, Substance Use Disorder, Psychotic Disorder, etc.).
3. Any medical condition that would contraindicate participation in deep breathing practices associated with relaxation training. Some examples may include, but are not limited to, increased intracranial pressure, unstable head or neck injury, active hemorrhage, recent spinal injury, empyema, bronchopleural fistula, flail chest, uncontrolled hypertension, anticoagulation, rib or vertebral fractures or osteoporosis, acute asthma or tuberculosis, recent heart attack, recent skin grafts in chest area, spinal fusions, bony metastases, brittle bones, bronchial hemorrhage, emphysema, untreated pneumothorax, and chest tubes.
4. Any history of epileptic seizure activity which may be worsened by prolonged exposure to a computer screen.
5. Participant is unable to hold small object between thumb and forefinger.
6. Participant is unable to manipulate computer keyboard or computer mouse.
7. Participant has substantial visual deficit in both eyes, which cannot be corrected, that would interfere with ability view a small screen on a mobile device or a laptop screen.
8. Participant is unable to wear a cheststrap heart monitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-15 (Estimated); Primary Completion 2019-07-15 (Estimated); Study Completion 2019-07-15 (Estimated)

PRIMARY OUTCOMES:
Anxiety Disorders Interview Schedule - 5 (ADIS-5) | Baseline, post-treatment change in outcome 4 days after session 8, and follow-up change in outcome 6-weeks after session 8.
  Diagnostic interview for anxiety disorders
Beck Anxiety Inventory | Baseline, post-treatment change in outcome 4 days after session 8, and follow-up change in outcome 6-weeks after session 8.
  21-item symptom checklist. Total score will be used as outcome. Total score ranges from 0-63, with higher scores indicating more anxiety.
COPE | Baseline, post-treatment change in outcome 4 days after session 8, and follow-up change in outcome 6-weeks after session 8.
  60-item measure assessing a broad range of coping responses. There are 15 subscales, each representing a different coping skill and each ranging in score from 4-16, with higher scores indicating more frequent usage of each of the 15 measured coping skills.
Perceived Stress Scale | Baseline, post-treatment change in outcome 4 days after session 8, and follow-up change in outcome 6-weeks after session 8.
  10-item measure of perceived stress. Total score used as primary outcomes. Total scores range from 0-40 with higher scores indicating higher levels of perceived stress.

SECONDARY OUTCOMES:
Functional outcome (sleep) | Baseline, post-treatment change in outcome 4 days after session 8, and follow-up change in outcome 6-weeks after session 8.
  Subject report of average hours of sleep per night

CONTACTS AND LOCATIONS:
Overall Officials: IRB Chairperson, Study Chair — East Tennessee State University

IPD SHARING:
Plan to Share IPD: No